CLINICAL TRIAL: NCT03617744
Title: Sleeve Gastrectomy for Morbid-Obesity Sequelae After Transplantation: A Randomized Controlled Trial Comparing Sleeve Gastrectomy Following Liver Transplantation to No Surgical Intervention in Patients With Morbid Obesity
Brief Title: Sleeve Gastrectomy for Morbid-Obesity Sequelae After Transplantation
Acronym: SG-4MOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-6286
Record Dates: First submitted 2018-06-04; First posted 2018-08-06 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Liver Transplantation; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to group a or group b
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Intervention (Experimental): Open Sleeve gastrectomy procedure will be performed immediately following liver transplantation (as a single surgery) or within 2 weeks of transplantation (as a second open surgery)
  Interventions: Procedure: Sleeve gastrectomy
- No Surgical Intervention (No Intervention): Liver transplantation will proceed as per routine practice

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Open sleeve gastrectomy
  Arms: Surgical Intervention

SUMMARY:
Complications associated with excess weight (hypertension, coronary artery disease and diabetes) have become major causes of morbidity and mortality after liver transplantation (LT). To ensure excellent long-term outcomes with LT it is critically important to understand the best strategies to minimize obesity and its associated complications in our patients. Weight loss can be achieved through dieting and exercise, but most patients are unable to maintain the weight loss. In the general population, bariatric surgery is much more effective than medical treatment for permanent weight loss and prevention or reduction of obesity-associated complications.

The purpose of this study is to determine the safety and effectiveness of performing sleeve gastrectomy (SG) procedure in the early post-LT period in obese patients.

The patient population for this study will be anyone listed for liver transplantation at Toronto General Hospital (University Health Network, Toronto, ON, Canada) and meeting the current standard criteria for bariatric surgery (BMI>40, or BMI>35 with at least 1 obesity-related complication).This study will randomly assign eligible participants to one of two groups (1:1). Patients in group 1 will receive standard lifestyle/diet counselling while patients in group 2 will undergo SG-specific counselling prior to transplant and the SG procedure within 2 weeks of LT (if safe to do so).

All participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* actively listed for liver transplantation at University Health Network
* BMI at screening of a) >40; or b) BMI >35 and 1 obesity-related complication [diabetes (defined as hyperglycemia requiring medication(s) for control), hypertension (defined as a persistently elevated systolic pressure greater than 140 mmHg and/or requiring medication(s) for control), hypercholesterolemia (defined as elevated lipids requiring medication for control)] OR a diagnosis of Non Alcoholic Fatty Liver Disease (defined as the presence of a fatty liver on imaging without a secondary cause such as alcohol abuse) or Non Alcoholic Steatohepatitis
* upper endoscopy showing no contraindications to a sleeve gastrectomy procedure

Exclusion Criteria:

* • Listed for re-transplantation, or transplantation of another organ (eg. kidney).

  * Previous bariatric surgery.
  * Contraindication to undergoing sleeve gastrectomy such as severe gastroesophageal reflux disease or Barrett's Esophagus
  * MELD (Model End-Stage Liver Disease) score > 35 at the time of transplantation
  * Presence of any condition that in the opinion of the investigator(s) could compromise the patient's ability to comply with study procedures
  * Patients with a BMI <32 at transplant or having weight loss of 20% or more (pre-transplant estimated dry body weight compared to estimated dry body weight at screening)
  * Presence of any other condition that, in the opinion of the investigator(s), could compromise the patient's ability to safely undergo, or benefit from, the SG procedure (eg. significant sarcopenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
morbid obesity | 12 months post-liver transplant
  rate of morbid obesity defined as BMI greater than or equal to 35

SECONDARY OUTCOMES:
mortality | 12 months post-transplant
  patient mortality
surgical morbidity | 12 months post-transplant
  rate of surgical morbidity
surgical morbidity | 3 months post-transplant
  rate of surgical morbidity
mortality | 3 months post-transplant
  patient mortality
change in weight | 12 months
  weight loss or gain as percentage of estimated "dry" weight at transplantation
surgical complications | 12 months
  rate of surgical complications
sleep apnea | 12 months post-transplantation
  percentage of participants in each group requiring BiPAP or CPAP for treatment of sleep apnea
hypertension | 12 months post-transplantation
  percentage of participants in each group requiring treatment of hypertension
diabetes | 12 months post-transplantation
  percentage of participants in each group requiring medical treatment of diabetes
hyperlipidemia | 12 months post-transplantation
  percentage of participants in each group requiring medical treatment of elevated lipids

CONTACTS AND LOCATIONS:
Overall Officials: David R Grant, M.D., Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No